CLINICAL TRIAL: NCT02558465
Title: Special Drug Use Investigation of Xarelto for VTE
Brief Title: Special Drug Use Investigation of Xarelto for Venous Thromboembolism (VTE)
Acronym: JPMS-XAR-VTE
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 17522; XAR-PE-DVT (Other: company internal)
Record Dates: First submitted 2015-09-23; First posted 2015-09-24 (Estimated); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Venous Thromboembolism
Keywords: Xarelto, rivaroxaban, VTE, PE, DVT, Japan, PMS, SDUI
MeSH Terms: conditions — Venous Thromboembolism; Venous Thrombosis | interventions — Rivaroxaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Rivaroxaban (Xarelto, BAY59-7939): Rivaroxavban administration group
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY59-7939) — Treatment parameters following the summary of product characteristics and the physician's decision

SUMMARY:
The objective of this investigation is to assess safety and effectiveness of Xarelto under practice routine use in VTE secondary prevention after acute DVT, focusing on hemorrhagic-related AEs, recurrent venous thromboembolism (PE/DVT), all-cause mortality. This study is a company sponsored, one- arm prospective cohort study with patients to whom Rivaroxaban treatment for VTE (PE/DVT) has been chosen. The study includes a standard observation period (1 year) and an extension survey period (2 years, at the longest).

ELIGIBILITY:
Inclusion Criteria:

- Patients who start rivaroxaban for VTE(pulmonary embolism, deep vein thrombosis) anticoagulation therapy.

Exclusion Criteria:

- Patients who are contraindicated based on the product label and have already received Xarelto treatment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Female and male patients who start rivaroxaban for VTE （pulmonary embolism, deep vein thrombosis) anticoagulation therapy
Sampling Method: Non-Probability Sample
Enrollment: 2540 (Actual)
Dates: Start 2015-11-13 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with ISTH (International Society on Thrombosis and Haemostasis) major bleeding as a measure of Safety and tolerability | Up to 2 years
Number of participants with symptomatic recurrent VTE (composite of DVT or nonfatal or fatal pulmonary embolism) | Up to 2 years

SECONDARY OUTCOMES:
Composite number of all-cause mortality, vascular events (acute coronary syndrome, ischemic stroke, transient ischemic attack, or systemic embolism), clinically relevant non-major bleeding and all other adverse events/ADRs | Up to 2 years
Number of participants with asymptomatic deterioration of thrombotic burden (change of D-dimer, imaging test such as CT or CCUS) by the end of standard observation period | at 1 year
Frequency of VTE recurrence and adverse events/ADRs comparison between distal and/or proximal DVT localization treatment outcomes | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many locations, Multiple Locations, Japan

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- [Derived] Fukuda I, Hirayama A, Kawasugi K, Kobayashi T, Maeda H, Nakamura M, Yamada N, Tajima T, Tachiiri M, Okayama Y, Sunaya T, Hirano K, Hayasaki T. Safety Profile and Effectiveness of Rivaroxaban for Patients With Venous Thromboembolism in Japan - Results From Post-Marketing Surveillance (XASSENT). Circ J. 2023 Aug 25;87(9):1175-1184. doi: 10.1253/circj.CJ-23-0104. Epub 2023 May 27. PMID 37245989
- See also: Click here to find information for studies related to Bayer products. To find this study enter the ClinicalTrials.gov identifier (NCT) number or Bayer Study Identifier (ID) in the search field. — http://clinicaltrials.bayer.com/